CLINICAL TRIAL: NCT04142281
Title: A Novel Estimation of Energy Balance Through the Calibration of Consumer Devices in Free-living, Rural US Children
Brief Title: ILSI Energy Balance Study
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: International Life Sciences Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 17030190
Record Dates: First submitted 2018-04-05; First posted 2019-10-29 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2019-10

CONDITIONS: Physical Activity
Keywords: Energy Balance; Metabolism
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Participants will provide a urine samples after which will be analyzed to calculate elimination rates of the doubly-labeled water isotopes from the body.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to apply measurement error techniques on consumer devices to assess rate of energy storage [ES] and energy expenditure [EE], then estimate EI using the intake-balance technique.

The goal of this study is to develop calibration models that will be able to be translated to other consumer devices with only minor modifications given common hardware (e.g. triaxial accelerometry), resulting in overall improved ability to assess energy balance and EI at a population level and positive health outcomes.

DETAILED DESCRIPTION:
There are four stages in the proposed project: 1) We will validate EE and ES (hereafter, Fitbit_EE and Fitbit_ES) from a consumer physical activity monitor (Fitbit Alta HR™) and body composition analyzer (Fitbit Aria™) with gold-standard measures of DLW for EE and DXA for ES during a 14-day baseline period; 2) We will estimate EI using the intake-balance method during the 14-day baseline period; 3) We will calibrate daily Fitbit_EE and Fitbit_ES from consumer devices using a Bayesian semi-parametric measurement error modeling approach to estimate energy balance; 4) We will reassess our validation and calibration models of consumer devices during a 14-day post-study assessment period to evaluate changes associated with growth and development with gold-standard measures of DLW for EE and DXA for ES.

Aims of the proposed study are to:

Specific Aim 1. Validate and calibrate consumer devices to estimate energy balance using gold-standard methods and a Bayesian semi-parametric approach. Hypothesis 1: We will be able to jointly model measurement error for both EE and ES to create a calibration model that reduces bias and improves accuracy of consumer devices of EE and ES.

Specific Aim 2. Estimate energy intake using the intake-balance technique using consumer monitors. Hypothesis 2:We will use calibrated EE and ES from consumer monitors to estimate EI using the intake-balance technique, with values being superior to self-reported EI.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children and adults, aged 8-90.
* Able to be physically active.

Exclusion Criteria:

* History of restrained eating, eating disorders, bariatric surgery, or other significant medical diagnosis that could impact metabolism.
* Participants taking thyroid medications, beta blockers, or other stimulants (medications are known to affect metabolism).

Ages: 8 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will include 24 children or adults, ages 8-90.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-01-13 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
Energy intake | 8 weeks
  Energy intake will be assessed subjectively via interviewer-administered dietary recalls. Three dietary recalls will occur on randomly selected non-consecutive days over each one-week treatment condition (including at least one weekend day) to minimize preparation that could bias recall by the participants. All interviews will be conducted over the telephone, will ask about all foods consumed over the previous 24 hours using a multi-pass approach, and energy intake will be calculated using the Nutrient Data System for Research software (NDSR Version 2014).

SECONDARY OUTCOMES:
Energy expenditure | 2 weeks
  Energy expenditure will be assessed using the doubly labelled water (DLW) technique over a two week period.
Body composition | 8 weeks
  Assessment of body composition, including fat mass, fat free mass, and visceral adipose tissue, will be completed using dual energy X-ray absorptiometry (DXA).

CONTACTS AND LOCATIONS:
Overall Officials: Robin Shook, PhD, Principal Investigator — Children's Mercy Kansas City
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT04142281/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT04142281/SAP_001.pdf